CLINICAL TRIAL: NCT04096287
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single-Ascending-Dose Trial to Evaluate the Safety, Tolerability, Immunogenicity, and Pharmacokinetics of Intravenous PNT001 in Healthy Volunteers
Brief Title: Safety and Tolerability of PNT001 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pinteon Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: PNT001-001
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PNT001 (Experimental): Single escalating doses of intravenous PNT001 administered as a 30 minute infusion at doses of 33mg, 100mg, 300mg, 900mg, 2700mg, and as a 60 minute infusion at 4000 mg
  Interventions: Biological: PNT001
- Placebo (Placebo Comparator): Single intravenous dose of vehicle administered as a 30 minute infusion up to 2700 mg and as a 60 minute infusion at 4000 mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: PNT001 — PNT001 diluted in 5% dextrose
  Arms: PNT001
Drug: Placebo — 5% dextrose
  Arms: Placebo

SUMMARY:
This first in human study is a multi-center, randomized, double-blind, placebo-controlled single ascending dose study to evaluate the safety, tolerability, pharmacokinetics, and immunogenicity of intravenous PNT001 in healthy adult participants.

DETAILED DESCRIPTION:
This Phase 1 clinical trial is a multicenter, double-blind, single ascending dose trial evaluating safety in up to a total of 48 participants across up to 6 dose cohorts, 5 planned and 1 to be determined if an additional dose group is required. Each cohort will include 8 participants (6 active, 2 placebo) who will receive a single dose of either PNT001 or placebo. Within each cohort a sentinel group of 2 participants (1 active, 1 placebo) will be enrolled to evaluate safety and tolerability before enrolling the full cohort. If there are no safety concerns (as determined by the data and safety monitoring board [DSMB]), the remaining 6 participants (randomized as 5 active, 1 placebo) will be enrolled. This process will be followed for all additional cohorts.

After screening, and laboratory assessments at Day -1, eligible participants will be admitted to the research unit on Day 1 (or Day -1 at Investigator's discretion), where they will remain for three (or four) nights with standardized meals provided during their inpatient stay. On Day 1, participants will be randomized to receive either active drug or placebo. Study medication will be administered as a single i.v. infusion over 30 minutes (up to 60 minutes for doses greater than 2,700 mg), followed by collection of safety, tolerability, and PK data over 16 weeks. Participants will be discharged on Day 4 and will return for an outpatient study visit on Day 5 (may be phone or clinic visit), and to the study site on Days 7, 14, 28, 42, 56, 70, 84, 98, and 112.

ELIGIBILITY:
Inclusion Criteria:

* The participant provides written informed consent.
* The participant is a male or female (not of childbearing potential), 21 to 65 years of age at time of screening.
* Female participants must have documented proof that they are not of childbearing potential and must not currently be breastfeeding.
* Male participants must agree to use barrier contraceptives plus spermicide and refrain from sperm donation during the entire study and for 200 days after dosing has been completed.
* The participant must not have participated in a clinical drug trial within 3 months of study start, or within 5 half-lives, unless the study blind has been broken and the participant was known to be on placebo
* The participant must have a body mass index of 18.5 to 30 kg/m^2

Exclusion Criteria:

* Any contraindication or inability to undergo lumbar puncture due to anticoagulant use, platelet level, or coagulation study/INR result
* Any significant acute or chronic medical illness
* Any history of cancer within 5 years of enrollment, with the exception of resected skin basal cell carcinoma
* Any major surgery within 4 weeks of study drug administration
* Donation of blood or serum > 500 mL to a blood bank or in a clinical study (except screening visit) within 3 months of study drug administration
* Inability to undergo venipuncture or tolerate venous access
* A history of smoking or using tobacco products within 3 months before study drug administration
* A history of drug or alcohol abuse as defined in DSM V, Diagnostic Criteria for Drug and Alcohol Abuse
* Evidence of any clinically significant neurological or psychiatric disorder that could interfere with study assessments as determined by investigator and sponsor
* A history or current status of schizophrenia, schizoaffective disorder or bipolar disorder, untreated major depression (DSM-V or ICD-10 criteria)
* Any significant illness or infection requiring intervention within the prior 30 days as determined by the investigator and sponsor
* An indication of potential suicidality risk based on the C-SSRS assessment
* Any of the following abnormalities:
* serum creatinine > 1.5 mg/dL at screening
* AST or ALT > 2x the upper limit of normal at screening
* blood pressure > 140/90 Hg at screening or baseline
* QTcF > 470 msec at screening or baseline
* A known hypersensitivity to any components of the PNT001 drug product or placebo (5% dextrose)
* Current use of or plan to use any medication (prescription or over-the-counter) that would potentially affect the assessment of the pharmacokinetics, pharmacodynamics, or immunogenicity of PNT001

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events | 16 weeks
  assess adverse events during 16 week duration of study
Incidence of Treatment Emergent Clinical Laboratory Test Abnormalities | 16 weeks
  measure clinical laboratory values during 16 week duration of study
Incidence of Treatment Emergent Abnormalities in Physical Examination Findings | 16 weeks
  observe skin, eyes, ears, nose, throat, cardiac and pulmonary status, abdomen, and extremities for any abnormalities
Incidence of Treatment Emergent Abnormalities in Neurological Examination Findings | 16 weeks
  perform a neurological assessment of orientation, cranial nerve function, limb function for presence of involuntary movements, muscle mass, tone, and strength, coordination, reflexes, sensation, joint position, gait, Romberg test
Incidence of Treatment Emergent Abnormalities in Blood Pressure | 16 weeks
  measure resting pulse rate as beats per minute
Incidence of Treatment Emergent Abnormalities in Pulse Rate | 16 weeks
  measure systolic and diastolic blood pressure in mmHg
Incidence of Treatment Emergent Abnormalities in 12 lead Electrocardiogram Assessment | 16 weeks
  measure QT and calculate QTcF value

SECONDARY OUTCOMES:
Pharmacokinetic properties of PNT001 in Serum | 16 weeks
  measure concentration of PNT001 in serum
Pharmacokinetic properties of PNT001 in Cerebrospinal Fluid (CSF) | 28 days
  measure concentration of PNT001 in CSF

OTHER OUTCOMES:
Pharmacodynamic effects of PNT001 in Cerebrospinal Fluid - total tau | 28 days
  measure CSF concentrations of total tau
Pharmacodynamic effects of PNT001 in Cerebrospinal Fluid - cis-pT231 tau | 28 days
  measure CSF concentrations of cis-pT231 tau
Pharmacodynamic effects of PNT001 in Cerebrospinal Fluid - total pT231 tau | 28 days
  measure CSF concentrations of total pT231 tau
Pharmacodynamic effects of PNT001 in Cerebrospinal Fluid - NfL | 28 days
  measure CSF concentrations of Neurofilament Light Chain (NfL)
Pharmacodynamic effects of PNT001 in Serum - NfL | 28 days
  measure serum concentrations of Neurofilament Light Chain (NfL)
Immunogenicity of PNT001 - ADA | 16 weeks
  measure presence of antidrug antibodies (ADA) in serum

CONTACTS AND LOCATIONS:
Overall Officials: Larry D. Altstiel, MD, PhD, Study Director — Pinteon Therapeutics, Inc
Locations (4):
- United States (4):
  - Woodland Research Northwest, Rogers, Arkansas
  - Pacific Research Network, Inc., San Diego, California
  - Hassman Research Institute, Marlton, New Jersey
  - Worldwide Clinical Trials, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No